CLINICAL TRIAL: NCT05293028
Title: Phase I Clinical Study of Safety, Tolerability, Preliminary Efficacy and Pharmacokinetics of F527 in the Treatment of Patients With Relapsed or Refractory Lymphoma
Brief Title: Study of F527 in Patients With Relapsed or Refractory Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTP-F527-001
Record Dates: First submitted 2022-03-03; First posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Relapsed/Refractory Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drug:F527 (Experimental): F527 is dose-escalated sequentially by accelerated titration and i3+3 design.
  Interventions: Drug: F527

INTERVENTIONS:
Drug: F527 — 0.001、0.01、0.1、0.3、1、3 and10 mg/kg QW

SUMMARY:
This study is a non-randomized, open-label, phase I dose-finding and dose-expansion study to evaluate the safety, tolerability, antitumor efficacy, PK and immunogen of F527 in patients with relapsed or refractory lymphoma sexual characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 and ≤80 years old;
2. Patients with histopathologically confirmed relapsed/refractory lymphoma; relapsed/refractory was defined as a patient who did not achieve a response (including complete or partial response) after the last systemic therapy regimen, or had disease progression after achieving a response or relapse;
3. Subjects must have at least one measurable lesion assessed by the investigator (long diameter of lymph node>15mm, long diameter of extranodal lesion>10mm);
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0-2;
5. Expected survival period ≥ 3 months;
6. The function of vital organs meets the following requirements (do not use any blood components and cytokines within 7 days before the first dose):

   Blood routine: neutrophil count ≥1.5×109/L; platelet count ≥75×109/L; hemoglobin ≥95g/L; Liver function: TBIL≤1.5×ULN, ALT and AST≤2.5×ULN; if there is liver metastasis, ALT and AST≤5×ULN; Renal function: creatinine≤1.5×ULN; Coagulation function: International Normalized Ratio (INR)≤1.5×ULN and Activated Partial Thromboplastin Time (APTT)≤1.5×ULN;
7. Understand the test procedures and content, and sign the informed consent voluntarily.

Exclusion Criteria:

1. Special types of lymphoma such as primary/secondary central nervous system lymphoma, etc.;
2. Patients with a history of other malignant tumors within the past 5 years, except for locally curable cancers (such as basal cell or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the prostate, cervix or breast, etc.);
3. History of hemolytic anemia or Evans syndrome in the last three months;
4. Positive direct antiglobulin test;
5. Those who have used CD47-targeted drugs or signal-regulated protein alpha (SIRPα)-targeted drugs in the past;
6. Received anti-tumor-related treatments such as anti-tumor chemotherapy, radiotherapy, biological therapy, or immunotherapy/immunomodulation therapy within 2 weeks before the first administration; the toxicity of previous anti-tumor therapy has not recovered to ≤ grade 1 (except for alopecia);
7. Patients who have a history of organ transplantation or allogeneic bone marrow transplantation, or who have received autologous stem cell transplantation within 3 months before the first administration or have other severe immunodeficiency;
8. HIV positive patients, syphilis-infected patients (RPR positive and TPPA positive) or active hepatitis (HBsAg positive and/or HBcAb positive, and HBV-DNA positive or higher than the upper limit of normal; HCV antibody positive and HCV- RNA positive or above the upper limit of normal);
9. Patients with uncontrollable or severe cardiovascular disease, who have New York Heart Association (NYHA) class II or above congestive heart failure, unstable angina, myocardial infarction and other cardiovascular diseases within 6 months before the first administration; Uncontrolled hypertension (systolic blood pressure ≥180mmHg and/or diastolic blood pressure ≥100mmHg);
10. Patients who have received any other clinical trial drug treatment within 4 weeks before the first dose;
11. Patients who have received live attenuated vaccine within 4 weeks before the first dose;
12. Patients who have a history of severe allergies, or who are known to be allergic to macromolecular protein preparations/monoclonal antibodies and any components of the investigational drug;
13. Patients with a history of mental illness or drug abuse;
14. Pregnant or lactating women, female patients or male patient partners who plan to become pregnant during the study period to 6 months after the last dose, and are reluctant to use a medically recognized effective contraceptive method (such as an intrauterine device or an intrauterine device) during the trial. condoms);
15. Patients who are judged by the investigator to be unsuitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2022-05-20 (Estimated); Primary Completion 2023-11-20 (Estimated); Study Completion 2024-05-20 (Estimated)

PRIMARY OUTCOMES:
DLTs | Up to 21 days
  Incidence of dose-limiting toxicities (DLTs) from the first dose through the end of the DLT observation period
Maximum Tolerated Dose (MTD) | Up to 21 days
  Maximum Tolerated Dose
RP2D | Up to 21 days
  PR2D will be determined by the sponsor and investigator based on the comprehensive data obtained on drug safety and tolerability, PK, preliminary anti-tumor efficacy, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China